CLINICAL TRIAL: NCT06964685
Title: Observational Assessment of Support With Impella® Best Practices in Acute Myocardial Infarction Complicated by Cardiogenic Shock
Brief Title: Assessment of Support With Impella® Best Practices in Acute Myocardial Infarction Complicated by Cardiogenic Shock
Acronym: OASIS-AMICS
Status: Recruiting | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ABMD-CIP-2024-04
Record Dates: First submitted 2025-04-07; First posted 2025-05-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: AMI Cardiogenic Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Impella — US commercially approved Impella CP is the device that study inclusion will be based on. Only patients with AMICS who receive Impella CP as the first Impella device after cardiogenic shock onset will be included in the study.

SUMMARY:
The observational study titled "Observational Assessment of Support with Impella Best Practices in Acute Myocardial Infarction Complicated by Cardiogenic Shock (OASIS-AMICS)" aims to evaluate the safety outcomes of patients with acute myocardial infarction complicated by cardiogenic shock (AMICS) who receive Impella CP during percutaneous coronary intervention (PCI) and who are managed with Impella best practices while receiving guideline-directed standard of care. This prospective, multicenter study will enroll up to 250 hemodynamically unstable patients with cardiogenic shock of less than 12 hours duration and acute myocardial infarction (AMI) of less than 24 hours duration. Cardiogenic shock will be confirmed by tissue hypoperfusion (lactate ≥ 2.5mmol/L and/or SvO2 <55% with a normal PaO2) and systolic blood pressure <100 mmHg and/or need for vasopressor therapy (dopamine/norepinepherine or epinephrine). Patients will be assessed for various safety endpoints, including a composite safety endpoint involving major bleeding, acute limb ischemia, and acute kidney injury. Secondary endpoints will evaluate all-cause mortality, major adverse cardiovascular and cerebrovascular events (MACCE), and hospitalizations through 1-year post-Impella implant. All patients presenting with AMICS at study sites will be screened for inclusion in the study after hospital discharge (or after death, if prior to hospital discharge). IRB approved consent waiver will be used to collect data from electronic health records from; Impella placement to discharge and post-discharge at 30 days post-Impella implant, 6 months post-Impella implant, and 1 year post-Impella implant.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction (AMI) of <36 hours duration from symptom onset to cath lab arrival, confirmed by:

  * ECG and/or biomarker evidence of ST-segment elevation myocardial infarction (STEMI) or
  * ECG and/or biomarker evidence of non-ST-segment elevation myocardial infarction (NSTEMI) and angiographic evidence of one or more culprit vessels
* Cardiogenic shock that develops under one of the following conditions: prior to primary PCI, with <24 hours from the onset of shock to cath lab arrival, or within 12 hours after initiating primary PCI. Cardiogenic shock is confirmed by at least two of the following:

  * Peripheral signs of tissue hypoperfusion (arterial blood lactate ≥2.5 mmol/l or SvO2 <55% with a normal PaO2)
  * Systolic blood pressure <100 mmHg or need for vasoactive agents to maintain systolic blood pressure ≥100 mmHg
  * Hemodynamic criteria represented by a cardiac index of <2.2 L/min/m2 or a cardiac power output ≤0.6 W
* Patient received PCI to treat the AMI
* Patient was supported with Impella CP as the initial MCS device for cardiogenic shock
* Age ≥18 years

Exclusion Criteria:

* Any contraindication listed in the Impella CP IFU if known to be present (i.e. mural thrombus in the left ventricle; presence of a mechanical aortic valve or heart constrictive device; aortic valve stenosis/calcification (equivalent to an orifice area of 0.6 cm2 or less); moderate to severe aortic insufficiency (echocardiographic assessment graded as ≥ +2); severe arterial disease precluding placement of the Impella system; presence of an atrial or ventricular septal defect (including post-infarct VSD); significant right heart failure; left ventricular rupture; cardiac tamponade; combined cardiorespiratory failure).
* 2. Shock principally due to a cause other than LV failure, including:

  * RV infarction, hypovolemia, anaphylaxis, hemorrhage, sepsis, myocarditis, pulmonary embolism, pneumothorax, or high cardiac output shock
  * Severe arrhythmias as the primary cause of low cardiac output
  * Known mechanical complications of AMI that may cause cardiogenic shock such as free wall rupture, ventricular septal defect or papillary muscle rupture with acute mitral regurgitation
* Other mechanical circulatory support already in place for present indication, including intra-aortic balloon counter-pulsation or patients with Impella CP placement prior to transfer to the cath lab at the tertiary facility
* Acute or chronic aortic dissection
* Prior PCI at another institution for the present infarction
* Thrombolytic therapy for the present infarction
* Not obeying verbal commands after preadmission or in-hospital cardiac arrest, indicative of possible anoxic brain injury NOTE:
* Non-intubated subjects: A positive and appropriate response to commands must be repeatable on at least two (2) instances to rule out reflex response to voice
* Intubated subjects: May be included if:

  * They were following verbal commands immediately prior to intubation, or
  * They were clearly following verbal commands after intubation
* Infective endocarditis
* Other severe, concomitant disease with limited life expectancy <1 year (other than cardiogenic shock)
* Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device that has not reached the timing of its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients with AMICS who receive Impella CP as the first Impella device after cardiogenic shock onset will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Composite Safety | All in-hospital events through discharge, an average of 15 days
  Composite safety endpoint (major bleeding, acute limb ischemia, or acute kidney injury requiring renal replacement therapy)

SECONDARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | Up to 1 year post-Impella implant
All-cause mortality | Up to 1 year post-Impella implant
Cardiovascular death | Up to 1 year post-Impella implant
Cardiovascular hospitalizations | Up to 1 year post-Impella implant
Heart failure hospitalizations | Up to 1 year post-Impella implant
Heart transplant or durable LVAD implantation | Up to 1 year post-Impella implant
Any new renal replacement therapy (RRT) | Up to 1 year post-Impella implant
Acute kidney injury (AKI) | In-hospital through discharge, up to 15 days
Major bleeding | In-hospital through discharge, up to 15 days
Hemolysis | In-hospital through discharge, up to 15 days
Acute limb ischemia (ALI) | In-hospital through discharge, up to 15 days
Major vascular complications | In-hospital through discharge, up to 15 days
Stroke | In-hospital through discharge, up to 15 days
Worsening Aortic Regurgitation | In-hospital through discharge, up to 15 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - St. Joseph Hospital Orange, Orange, California
  - Ascension via Christi, Wichita, Kansas
  - New Mexico Heart, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kapur NK, Kanwar M, Sinha SS, Thayer KL, Garan AR, Hernandez-Montfort J, Zhang Y, Li B, Baca P, Dieng F, Harwani NM, Abraham J, Hickey G, Nathan S, Wencker D, Hall S, Schwartzman A, Khalife W, Li S, Mahr C, Kim JH, Vorovich E, Whitehead EH, Blumer V, Burkhoff D. Criteria for Defining Stages of Cardiogenic Shock Severity. J Am Coll Cardiol. 2022 Jul 19;80(3):185-198. doi: 10.1016/j.jacc.2022.04.049. PMID 35835491
- [Background] Gornik HL, Aronow HD, Goodney PP, Arya S, Brewster LP, Byrd L, Chandra V, Drachman DE, Eaves JM, Ehrman JK, Evans JN, Getchius TSD, Gutierrez JA, Hawkins BM, Hess CN, Ho KJ, Jones WS, Kim ESH, Kinlay S, Kirksey L, Kohlman-Trigoboff D, Long CA, Pollak AW, Sabri SS, Sadwin LB, Secemsky EA, Serhal M, Shishehbor MH, Treat-Jacobson D, Wilkins LR; Peer Review Committee Members. 2024 ACC/AHA/AACVPR/APMA/ABC/SCAI/SVM/SVN/SVS/SIR/VESS Guideline for the Management of Lower Extremity Peripheral Artery Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2024 Jun 11;149(24):e1313-e1410. doi: 10.1161/CIR.0000000000001251. Epub 2024 May 14. PMID 38743805
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Moussa ID, Klein LW, Shah B, Mehran R, Mack MJ, Brilakis ES, Reilly JP, Zoghbi G, Holper E, Stone GW; Society for Cardiovascular Angiography and Interventions. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Society for Cardiovascular Angiography and Interventions (SCAI). Catheter Cardiovasc Interv. 2014 Jan 1;83(1):27-36. doi: 10.1002/ccd.25135. Epub 2013 Oct 16. PMID 23894025
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511